CLINICAL TRIAL: NCT00482248
Title: An Open-label Extension Study to Assess Long Term Safety and Tolerability of Omalizumab Treatment in Adults and Adolescents With Severe Allergic Asthma Who Participated in the 52 Week CIGE250011E2 Study
Brief Title: Safety and Tolerability of Omalizumab in Adults and Adolescents With Severe Allergic Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIGE0250011E3
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: Asthma; anti-immunoglobulin E; omalizumab; allergic asthma
MeSH Terms: conditions — Asthma | interventions — Omalizumab

INTERVENTIONS:
Drug: Omalizumab

SUMMARY:
This study will assess further the safety and tolerability of long-term treatment with omalizumab by extending omalizumab treatment by 1 year for those patients with allergic asthma who successfully completed study CIGE25011E2.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of severe allergic asthma who completed the treatment period of CIGE250011E3 protocol, without experiencing any significant drug-related adverse events
* Male or female patients 12-75 years of age who have given written informed consent approved by the ethical committee

Exclusion Criteria:

* Patients who had not received study medication for greater than 84 days since visit 38 of study CIGE240011E3
* Pregnant females or nursing mothers
* Patients with know hypersensitivity to any ingredients of Omalizumab or related drugs

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 12 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2003-06; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Safety assessed by adverse events, serious adverse events, hematology, blood chemistry and urinalysis value, vital signs data, the performance of physical examinations and body weight measurements.

SECONDARY OUTCOMES:
Efficacy assessed by changes in forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC), the investigator's assessment of asthma control, corticosteroid use, the incidence of hospitalization and outpatients visits, and absenteeism fr

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals